CLINICAL TRIAL: NCT04905186
Title: The Effects of Different Domains of Executive Function Dual Task Walking on Brain Activation and Gait Performance in Healthy Adults
Brief Title: Different Domains of Executive Function Dual Task Walking on Brain Activation and Gait Performance in Healthy Adults
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202103125RINC
Record Dates: First submitted 2021-05-13; First posted 2021-05-27 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Executive Function; Neurosciences
Keywords: executive function; dual task walking; difficulty level; brain activity; motor performance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy adults: This is a cross-over study with no intervention.

SUMMARY:
The aim of this study is to investigate the effects of different domains of executive function (EF) during dual task walking condition on brain activation and gait performance in healthy adults. There are two experiments will be conducted in this study. Experiment 1 is a pilot study to determine the same level of difficulty in 3 EF domains, including inhibition, working memory and cognitive flexibility. Experiment 2 is carried out to investigate the effects of 3 different domains of EF which difficulties are controlled on gait performance and brain activation in dual task condition. 10 subjects will perform Stroop test (2s/3s/4s to change question), backward digit spans (3/4/5 digits) and naming test in Experiment 1. In Experiment 1, the primary outcome is the correct response speed (CRS) while secondary outcome will be the brain activity. In Experiment 2, 30 subjects will perform the single cognitive task A (SCTA, Stroop test), single cognitive task B (SCTB, backward digit spans), single cognitive task C (SCTC, naming test), single walking task (SWT), dual task A (DTA, walking while performing cognitive task A), dual task B (DTB, walking while performing cognitive task B) and dual task C (DTC, walking while performing cognitive task C). The CRS, gait performance, brain activity and the dual task costs (DTC) will be recorded in the Experiment 2. Brain activities in prefrontal cortex (PFC), premotor cortex (PMC) and supplementary motor area (SMAs) will be measured by functional near-infrared spectroscopy (fNIRS) during this study. One-way ANOVA with Tukey post-hoc test will be performed to establish the effect of different type of executive task on CRS or the brain activity. The differences of gait parameters and brain activity in different condition in the Experiment 2 will be examined by one-way ANOVA with repeated measured. Furthermore, the Pearson correlation coefficient will be used to examine the correlation of brain activation and executive function performance or gait parameters.

ELIGIBILITY:
Inclusion Criteria:

* 20-30 years (Experiment 1 & 2)
* Mini-Mental State Examination (MMSE) score greater than 24 points (Experiment 1 & 2)
* ability to walk 10 meters independently without an assistive device (Experiment 2)

Exclusion Criteria:

* any neurologic, orthopedic or psychological diseases (Experiment 1 & 2)
* color vision deficiency (Experiment 1 & 2)
* had the fall experiences within 6 months before the study (Experiment 2)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population in this study are heathy adults.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Experiment 1: Executive function performance- correct response speed (CRS) | Day 1
  CRS is the number of correct responses per unit time (correct responses/ second)
Experiment 2: Executive function performance- correct response speed (CRS) | Day 1
  CRS is the number of correct responses per unit time (correct responses/ second)
Experiment 2: walking performance- gait speed | Day 1
  The unit is m/s
Experiment 2: walking performance- cadence | Day 1
  The unit is steps/min
Experiment 2: walking performance- stride length | Day 1
  The unit is m
Experiment 2: dual task performance- dual task costs(DTC) in mobility | Day 1
  DTC in mobility = (single task gait speed - dual task gait speed) / single task gait speed x 100%
Experiment 2: dual task performance- dual task costs(DTC) in executive function | Day 1
  DTC in executive function = (single task correct response speed - dual task correct response speed) / single task correct response speed x 100%
Experiment 2: dual task performance- combine mean of dual task costs(DTC) | Day 1
  combine mean of DTC = ( DTC in mobility + DTC in executive function) / 2

SECONDARY OUTCOMES:
Experiment 1: Brain activation over prefrontal cortex | Day 1
  The unit is micro mole (μmol). A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics, including oxygenated-hemoglobin and de-oxygenated hemoglobin.
Experiment 1: Brain activities over supplementary motor area | Day 1
  The unit is micro mole (μmol). A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics, including oxygenated-hemoglobin and de-oxygenated hemoglobin.
Experiment 1: Brain activities over premotor cortex | Day 1
  The unit is micro mole (μmol). A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics, including oxygenated-hemoglobin and de-oxygenated hemoglobin.
Questionnaire in Chinese version | Day 1
  used for the participants to sort the task by the difficulty level based on their own experiences.The participants will be asked to grade the tasks from 1-10 scale. Scale one is the simplest and 10 is the hardest.
Experiment 2: Brain activities over prefrontal cortex | Day 1
  The unit is micro mole (μmol). A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics, including oxygenated-hemoglobin and de-oxygenated hemoglobin.
Experiment 2: Brain activities over supplementary motor area | Day 1
  The unit is micro mole (μmol). A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics, including oxygenated-hemoglobin and de-oxygenated hemoglobin.
Experiment 2: Brain activities over premotor cortex | Day 1
  The unit is micro mole (μmol). A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics, including oxygenated-hemoglobin and de-oxygenated hemoglobin.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan